CLINICAL TRIAL: NCT03924804
Title: Effect of Different Infusion Volume on Perioperative Bladder and Blood Volume in Patients Undergoing Daytime Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, Principal Investigator, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20190418
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Cholecystolithiasis and Thyroid Nodule
MeSH Terms: conditions — Cholecystolithiasis; Thyroid Nodule | interventions — Ringer's Solution

STUDY DESIGN:
Intervention Model Description: Doppler Ultrasonography Assessed Bladder and Blood Volume
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: 2 ml/kg group (Experimental)
  Interventions: Drug: Ringer's solution acetate
- Group B: 8 ml/kg group (Experimental)
  Interventions: Drug: Ringer's solution acetate
- Group C: 16 ml/kg group (Experimental)
  Interventions: Drug: Ringer's solution acetate

INTERVENTIONS:
Drug: Ringer's solution acetate — Intravenous infusion of 2 ml/kg Ringer's solution acetate within 1 hour after induction.
  Arms: Group A: 2 ml/kg group
Drug: Ringer's solution acetate — Intravenous infusion of 8ml/kg Ringer's solution acetate within 1 hour after induction.
  Arms: Group B: 8 ml/kg group
Drug: Ringer's solution acetate — Intravenous infusion of 16ml/kg Ringer's solution acetate within 1 hour after induction.
  Arms: Group C: 16 ml/kg group

SUMMARY:
The objective of the trial was to explore the effect of different infusion volume on perioperative bladder and blood volume in patients undergoing daytime surgery assisted by bladder and vascular ultrasound and transthoracic echocardiography.

DETAILED DESCRIPTION:
The objective of the trial was to evaluate the effects of different infusion volume of Ringer's solution acetate (2 ml/kg,8ml/kg, 16ml/kg) on bladder volume, hemodynamics,transthoracic echocardiography and vascular ultrasound including the inferior vena cava(IVC) and the right subclavian vein(SCV) diameter and the IVC and SCV collapsibility index in patients undergoing daytime surgery through a randomized controlled clinical study, so as to provide better guidance for clinical transfusion avoiding bladder catheterization . The patients in this trial were visited before induction and discharge from the postanaesthesia .We also collected the first time and times of micturition and whether the patients have the dysuria.

ELIGIBILITY:
Inclusion Criteria:

* 1. ethnic Chinese;
* 2. age, 18 to 65 years old;
* 3. American Society of Anaesthesiologists (ASA) physical status I or II;
* 4. Daytime patients scheduled for general anesthesia

Exclusion Criteria:

* Patients unwilling to cooperate with the experiment
* Body mass index exceeding 30 kg/m2;
* Patients with a history of heart ,liver and Renal failure ,hypertension,diabetes mellitus or arteriosclerosis; and any allergy to drugs used in the study.
* Patients with the urinary diseases, such as kidney, ureteral calculi and tumors, prostatic hypertrophy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
1. The change of bladder volume | baseline and 10 minutes before leaving the post-anesthesia care unite
  bladder and blood volume in patients undergoing daytime surgery assisted by bladder and vascular ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China